CLINICAL TRIAL: NCT04648319
Title: A Pilot Study of BMS-936558 With Stereotactic Ablative Radiation Therapy After Induction Chemotherapy in Cholangiocarcinoma
Brief Title: A Study of BMS-936558 With SBRT After Induction Chemotherapy in Cholangiocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: pharma company decision to withdraw the financial and IMP support
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIO-2019-0447; CA209-7DJ (Other Grant/Funding Number: CA209-7DJ)
Record Dates: First submitted 2020-11-11; First posted 2020-12-01 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2020-11

CONDITIONS: Cholangiocarcinoma
Keywords: cholangiocarcinoma; Immunotherapy; SBRT; PFS
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: single group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- locally advanced, metastatic or recurrent cholangiocarcinoma (Experimental): D1: Compound: BMS-936558 treatment d8: radiotherapy D 20: CT guided Biopsy D 28: BMS-936558 treatment monthly: BMS-936558 treatment CT CAP: after 4doses
  Interventions: Drug: BMS-936558

INTERVENTIONS:
Drug: BMS-936558 — BMS-936558 followed by 30 grays of 3 to 5 fractions of high dose SBRT followed by monthly BMS-936558 until progression
  Other Names: radiation therapy : SBRT

SUMMARY:
This is an Open-label, single-arm, multicenter Phase II pilot study to assess the efficacy and safety of BMS-936558 with stereotactic ablative radiation therapy after induction chemotherapy in cholangiocarcinoma.

DETAILED DESCRIPTION:
The current standard regimen for advanced biliary tract cancers as per NCCN guidelines (version 2.2019) is gemcitabine plus cisplatin. However, since no single chemotherapy agent or combination regimen has consistently led to durable tumor regression, prevention of recurrent obstruction following palliative intervention, and extension of survival beyond 8 to 15 months, there is a pressing need for new treatment approaches in patients with dismal prognosis. Recent discoveries in tumor immunology, paralleled by technological advances in radiation therapy, have provided promising role for combining ablative radiotherapy with targeted immune modulators (El Chediak et al., 2017).

objectives: Primary: To evaluate the progression-free survival (PFS) at 8 months and the disease control rate (DCR) in patients with non-resectable locally-advanced or metastatic or recurrent intrahepatic or extrahepatic cholangiocarcinoma (CCA) following BMS-936558 /stereotactic ablative radiation therapy (SBRT) treatment.

Secondary:

1) To evaluate the overall survival (OS) rate in patients with advanced intrahepatic or extrahepatic CCA following BMS-936558/SBRT treatment. .

3) To evaluate tumor response rates at the primary and secondary sites using the response evaluation criteria in solid tumors (RECIST1.1) criteria.

4) To evaluate the duration of response at non-irradiated tumor sites in patients with Stage IV disease.

5) To evaluate the following biomarkers: CD3+, CD4+, and CD8+ T cell infiltration, and changes in PD-L1 expression at baseline and following first cycle of BMS-936558 and SBRT.

6) To assess the safety and tolerability of BMS-936558/SBRT according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAEv5).

7) To assess the quality of life of the patients through completed FACT-Hep questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. Signed and dated informed consent form.
  2. Patients aged ≥18 years.
  3. Pathologically (histologically or cytologically) and radiologically confirmed diagnosis of non-resectable locally advanced or metastatic or recurrent intrahepatic or extrahepatic CCA within 90 days of registration.
  4. Patients who have stable disease or partial response following 4 cycles of cisplatin/gemcitabine.
  5. ECOG performance score <3

     o An estimated life expectancy of more than 3 months.
  6. Have adequate hematologic and biochemical function by meeting the following:

     * Total bilirubin acceptable level ≤ 1.5 × the institutional upper limit of normal (ULN) range;
     * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) acceptable levels up to 5 x ULN range;
     * Serum urea and serum creatinine acceptable levels up to 1.5 x ULN range;
     * Calculated glomerular filtration rate ≥ 45 mL/min according to the Chronic Kidney Disease Epidemiology Collaboration equation (or local institutional standard method).
  7. Negative serum or urine pregnancy test at screening for women of childbearing potential who are sexually active.
  8. Highly effective contraception for both males and females of child-bearing potential who are sexually active throughout the study and for at least 5 months and 7 months after the last BMS-936558 treatment administration, respectively.
  9. Candidate for percutaneous biopsy as per tumor location evidenced by CT scan and interventional radiologist.

Exclusion Criteria:

1. Patients who have progression following 4 cycles of cisplatin/gemcitabine evidenced by CT scan as per RECIST 1.1.
2. Active brain metastases or leptomeningeal metastases.
3. Prior organ transplantation or allogenic stem-cell transplantation.
4. Known prior severe hypersensitivity to IMP or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI-CTCAE v4.03 Grade ≥ 3).
5. Active infection requiring systemic therapy within 28 days before the first dose of study treatment (e.g., urinary tract infection).
6. Known history of testing positive for the human immunodeficiency virus or known acquired immunodeficiency syndrome.
7. Evidence of liver cirrhosis.
8. Current use of immunosuppressive medication, except for the following:

   * Intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection);
   * Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent;
   * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
9. Active autoimmune diseases that might deteriorate upon receiving an immune-stimulatory agent.
10. Conditions such as vitiligo, psoriasis, diabetes type I, or hypo- or hyper-thyroid diseases not requiring immunosuppressive treatment are eligible.
11. Commonly excluded conditions include: Addison's disease, thyroiditis/Hashimoto's thyroiditis, systemic lupus erythematosus, Sjogren's syndrome, scleroderma, myasthenia gravis, Goodpasture's syndrome, and Grave's disease
12. Hepatic insufficiency manifesting as clinical jaundice, hepatic encephalopathy, and/or variceal bleed within 60 days prior to study entry.
13. Transmural myocardial infarction within 6 months of enrollment; provided that anti-platelets cannot be stopped to perform percutaneous biopsy.
14. Congestive heart failure (≥ New York Heart Association Classification Class II) requiring hospitalization within the last 6 months provided that anti-platelets cannot be stopped to perform percutaneous biopsy.
15. Serious cardiac arrhythmia requiring medical treatment provided that anti-platelets cannot be stopped to perform percutaneous biopsy.
16. Recent cerebral vascular accident/stroke within 6 months of enrollment provided that anti-platelets cannot be stopped to perform percutaneous biopsy.
17. End-stage renal disease requiring dialysis.
18. Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis, or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior.
19. Vaccination within 4 weeks of the first dose of BMS-936558 and while on trial is prohibited except for administration of inactivated vaccines.
20. Treatment with an investigational agent within 28 days before the first dose of study treatment.
21. Prior treatment with any drug or antibody (anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody) targeting T cell co-stimulation or checkpoint pathways.
22. Patients suspected by the physician that he/she will not be compliant to the protocol conduct.
23. Pregnant women are excluded from this study; breastfeeding should be discontinued.
24. Patients participating in another clinical trial.
25. Patients not willing to sign the consent form.
26. Any psychiatric condition that would prohibit the understanding or rendering of informed consent.
27. Legal incapacity or limited legal capacity patients receiving other oncology specific medication not authorized in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
To evaluate the progression-free survival (PFS) at 8 months and the disease control rate (DCR) in patients with non-resectable locally-advanced or metastatic or recurrent intrahepatic or extrahepatic CCA following BMS-936558/SBRT treatment | 8 months
  will be done at 8 months of the initial patient diagnosis and after 8 cycles of treatment

SECONDARY OUTCOMES:
To evaluate the overall survival (OS) rate in patients with advanced intrahepatic or extrahepatic CCA following BMS-936558/SBRT treatment. | up to 2 years
  survival status will be evaluated every 3 months after progression
To evaluate tumor response rates at the primary and secondary sites using the response evaluation criteria in solid tumors (RECIST1.1) criteria. | every 4 months from the date of first treatment visit until the date of first documented progression, assessed up to 2 years.
  evaluation will be done by CT scan of chest ,abdomen and pelvis every 4 months from the D1 ( after each 4 cycles of treatment until progression )
To evaluate the duration of response at non-irradiated tumor sites in patients with Stage IV disease. | every 4 months from the date of first treatment visit until the date of first documented progression, assessed up to 2 years.
  evaluation will be done by CT scan of abdomen, pelvis and chest every 4 months (after every 4 cycles of treatment until progression )
To evaluate the following biomarkers: CD3+, CD4+, and CD8+ , and changes in PD-L1 expression at baseline and following first cycle of BMS-936558and SBRT. | at baseline/inclusion visit and Day20 (after radiotherapy)
  biomarkers will be assessed from baseline biopsy and after receiving first BMS-936558and SBRT for changes.
  CD3+, CD4+, and CD8+: Will be quantified in mm2 in the most abundant tumor-infiltrating area in both, the stroma and the tumor, of the baseline biopsy (continuous variable) PD-L1: Will be evaluated on tumor cells and infiltrating immune T cells and be classified as negative or positive or not applicable (categorical variable)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Shamseddine, MD, Principal Investigator — American University of Beirut Medical Center
Locations (4):
- Belgium (2):
  - Institut Jule Bordet, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
- American University of Beirut Medical Center, Beirut, Lebanon
- Centre hospitalier de Luxembourg, Luxembourg, Luxembourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elias C, Zeidan YH, Bouferraa Y, Mukherji D, Temraz S, Charafeddine M, Al Darazi M, Shamseddine A. A phase II single arm study of Nivolumab with stereotactic Ablative radiation Therapy after induction chemotherapy in CHOlangiocarcinoma (NATCHO). BMC Cancer. 2022 Dec 12;22(1):1296. doi: 10.1186/s12885-022-10373-1. PMID 36503610